CLINICAL TRIAL: NCT06630611
Title: Phase II Randomized Study Evaluating a Pragmatic Approach to Adoptive Cell Therapy (ACT) Using an IL2 Analog (ANV419) vs High Dose IL2 After Tumor Infiltrating Lymphocytes (TIL) Therapy in Patients With Melanoma, NSCLC and Cervical Cancer
Brief Title: Evaluation of a Pragmatic Approach to Adoptive Cell Therapy (ACT) Using an IL2 Analog (ANV419) vs High Dose IL2 After Tumor Infiltrating Lymphocytes (TIL) Therapy in Patients With Melanoma, NSCLC and Cervical Cancer (PragmaTIL)
Acronym: PragmaTIL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vall d'Hebron Institute of Oncology (Other)
Collaborators: Banc de Sang i Teixits (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VHIO23002
Record Dates: First submitted 2024-07-26; First posted 2024-10-08 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Melanoma; Non Small Cell Lung Cancer; Cervical Cancer
Keywords: Immune checkpoint blockade (ICB) resistant tumors; Tumor-Infiltrating Lymphocyte; Adoptive Cell Therapy; Interleukin-2 (IL-2)
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Uterine Cervical Neoplasms | interventions — Cyclophosphamide; fludarabine; Interleukin-2

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 over the two study arms. Randomization will be stratified by cancer type (melanoma and non-melanoma) and center following a block randomization. Of the total 40 patients, the first 10 patients recruited in the study will be metastatic melanoma patients. Of the remaining 30 patients 10 of them must be melanoma patients (20 in total) and the other 20 patients will be preferably NSCLC or cervical cancer, but additional patients with melanoma can also be included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Arm A) (Active Comparator): Patients will receive standard high dose of IL2 (HD-IL-2) after receiving standard lymphodepleting chemotherapy and TIL product. In the control arm, the first i.v. dose of HD-IL2 will be administered within 3-24 hours after TIL infusion, and thereafter every 8 hours to tolerance up to a maximum of 6 doses.
  Interventions: Biological: NMA-LD regimen; Biological: Tumor infiltrating lymphocytes adoptive cell therapy (TIL-ACT) infusion; Biological: High dose IL-2
- Experimental Arm (Arm B) (Experimental): Patients will receive IL2 analog (ANV419) after receiving standard lymphodepleting chemotherapy and TIL product. In the experimental arm, ANV419 (one dose) will be administered within 3-24 hours after TIL infusion.
  Interventions: Biological: NMA-LD regimen; Biological: Tumor infiltrating lymphocytes adoptive cell therapy (TIL-ACT) infusion; Biological: IL-2 analog

INTERVENTIONS:
Biological: NMA-LD regimen — The use of the NMA-LD regimen (cyclophosphamide and fludarabine) prior to cell administration is expected to lead to myelosuppression in all patients.
  Other Names: Cyclophosphamide and Fludarabine
Biological: Tumor infiltrating lymphocytes adoptive cell therapy (TIL-ACT) infusion — On Day 0 (at least 24h after the last dose of fludarabine) patients will be hospitalized in a dedicated unit. Autologous TIL infusion will be administered intravenously.
Biological: High dose IL-2 — Only for patients in Arm A.
  IL-2 begins between 3 and 24 hours after the completion of the TIL infusion and is given as a bolus administration every eight hours (minimum interval) to 24 hours (maximum interval) with a maximum of six doses from the beginning of each administration.
  Arms: Control Arm (Arm A)
Biological: IL-2 analog — Only for patients in Arm B
  ANV419 will be administered between 3 and 24 hours after the completion of the TIL infusion with a slow IV infusion over 15-30 minutes + 5 minutes once, at 243µg/kg.
  Arms: Experimental Arm (Arm B)

SUMMARY:
Background:

The presence of T-lymphocytes in resected tumor samples derived from long-term survival patients and the fact that reinvigoration of their functionality through the administration of specific immune-therapies can lead to remarkable antitumor responses supports that lymphocytes play a critical role in cancer immunity.

TIL-based ACT (Adoptive cell therapy using tumor-infiltrating lymphocytes product) is a modality of ACT used to treat patients with multiple types of cancer and it consists in the adoptive transfer of ex vivo expanded autologous tumor-infiltrating lymphocytes obtained from tumor resection or tumor biopsies in patients following a non-myeloablative lymphodepleting (NMA-LD) chemotherapy. Ex vivo expansion of TIL relies on the non-specific expansion of lymphocytes present in tumor single cell suspensions or tumor fragments in high dose IL-2.

Although proven efficacy in selected, the HD-IL-2 use remains relatively restricted due to toxicity. Due to the short serum half-life and the need to achieve an immune-modulatory effect in the tissues, IL-2 must be given in doses that induce severe systemic toxicities, including capillary leak syndrome (CLS), pulmonary edema, hypotension, acute renal insufficiency, and rarely myocarditis, limiting its applicability in cancer. Studies comparing HD-IL-2 with lower doses both in renal cell carcinoma and metastatic melanoma to minimize toxicity demonstrated the superiority of the high dose regimens in both diseases. These drawbacks of HD-IL-2 use encouraged the development of improved IL-2-based biologic agents with higher selectivity for effector immune cell subsets, reduced toxicity, and prolonged half-life.

ANV419 is a novel IL-2 agent, which has been developed as a preferentially IL-2Rβγ directed fusion protein with a longer half-life. It has shown high effector selectivity and a favorable safety profile in preclinical testing, including in nonhuman primates, and it has been investigated in an ongoing open-label, dose-escalation Phase I Study in multiple tumor types. he safety profile of ANV419 is characterized by pyrexia, nausea, vomiting, ALT/AST changes and CRS in some patients. Most events are low grade and self-limiting and manageable with standard supportive care. ANV419 was well-tolerated by most patients. No patient discontinued treatment due to treatment related AE.

Taking all the previous information into account, the primary objectives of this study are:

1. To determine whether TIL-ACT using the IL-2 analog ANV419 reduces the mean number of predefined grade ≥3 relevant adverse events related to interleukin use (based on Common Terminology Criteria for Adverse Events v5.0 - CTCAE v5.0) compared to TIL-ACT using HD-IL-2.
2. To determine whether TIL-ACT using the IL-2 analog improves patient´s reported outcomes (PRO) compared to TIL-ACT using HD-IL-2

DETAILED DESCRIPTION:
This is a an open-label, randomized, pragmatic multicenter phase II clinical trial to compare the safety, quality of life and efficacy of current protocols of adoptive cell therapy based on tumorinfiltrating lymphocytes (TIL-ACT) established at each institution facility through the randomization between two types of following interleukin used for engrafting and in vivo expansion of TILs: standard high-dose (HD) IL-2(600.000 IU/kg) or ANV419.

Total number of patients included in the trial will be 40. Of the total 40 patients, the first 10 patients recruited in the study will be metastatic melanoma patients. The melanoma and non-melanoma cohorts will be equally distributed between the two arms. Patients will be randomized to start treatment with either HD-IL-2 (Control arm) or with ANV419 (Experimental arm).

The objectives of this study are the following:

Primary objectives:

* To determine whether TIL-ACT using the IL-2 analog ANV419 reduces the mean number of predefined grade ≥3 relevant adverse events related to interleukin use (based on Common Terminology Criteria for Adverse Events v5.0 - CTCAE v5.0) compared to TIL-ACT using HD-IL-2.
* To determine whether TIL-ACT using the IL-2 analog improves patient´s reported outcomes (PRO) compared to TIL-ACT using HD-IL-2

Secondary objectives:

* To evaluate the safety and the tolerability of TIL-ACT using the IL-2 analog ANV419 compared to TIL-ACT using HD-IL-2.
* To evaluate short-term efficacy outcomes in patients receiving the IL-2 analog ANV419 or HD-IL-2.
* To evaluate long-term efficacy outcomes in patients receiving the IL-2 analog ANV419 or HD-IL-2.
* To evaluate the quality of life (QoL) and symptomatology in patients receiving the IL-2 analog ANV419 or HD-IL-2.
* To evaluate anxiety and depression in patients receiving the IL-2 analog ANV419 or HD-IL-2.
* To develop the health technology assessment (HTA) of TIL-ACT using ANV419, via the analysis of cost-effectiveness, budget impact, reimbursement strategies, user acceptance, and technical feasibility. This assessment, together with a social return of investment (SROI) analysis, will provide relevant information to participant member states regarding the possibility of implementing optimized and affordable treatments in their healthcare systems.

Exploratory objectives:

* To evaluate the impact of the different cytokine regimens on CD8+, NK and Treg proliferation, cytokine secretion profile, as well as the persistence and transcriptomic/phenotypic profile of the infused TIL product at different times following TIL infusion.
* To correlate the presence and persistence of tumor- and neoantigen- reactive TIL and their transcriptomic/phenotypic profile with clinical outcome.
* To evaluate the influence of tumor and neoantigen heterogeneity measured through tumor and cell free DNA sequencing prior to and during treatment.
* To evaluate biometric physiological parameters (mobility, heart rate, SpO2 and sleep cycle) through wearable devices during and after treatmen

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically proven metastatic or unresectable cutaneous melanoma, NSCLC, or cervical cancer. The disease must have progressed to at least one standard systemic anticancer therapy, regardless whether in the adjuvant or metastatic setting, or the patient is unable/unwilling to receive standard therapy. Patients who are receiving an anticancer treatment post-progression are also eligible to be included, at the investigator's discretion, always respecting the wash-out period for starting NMA-LD chemotherapy.
2. Patients must have at least one adequate lesion (primary tumor or metastasis) for resection or biopsy (with minimal morbidity, preferentially using imaging-guided minimally invasive procedures) for TIL generation.

   Note: If this lesion was previously irradiated, the lesion must have demonstrated progression prior to resection/biopsy.
3. Patients must have a remaining measurable disease as defined by RECIST v. 1.1 criteria following tumor resection/biopsy for TIL manufacturing.

   Note: Lesions previously irradiated should not be selected as target lesions unless there has been demonstrated progression in those lesions.
4. Patient must be at least 18 years old at the tissue procurement visit.
5. Patient must understand and voluntarily sign an informed consent document before any study-related assessments/procedures being conducted.
6. Patient must be able and willing to comply to the study visit schedule and protocol requirements.
7. Patients must have a clinical performance of Eastern Cooperative Oncology Group 0 or 1.
8. Patients are considered medically fit enough to undergo all study procedures and interventions and adequate hematological, renal, and hepatic functions defined by:

   1. Haemoglobin ≥9.0 g/dL.
   2. An absolute neutrophil count ≥ 1.5x10E9/L without the support of filgrastim.
   3. Platelets ≥100x10E9/L.
   4. PT and aPTT ≤1.5 x ULN (unless receiving therapeutic anticoagulation).

      - subjects receiving therapeutic anticoagulation (such as low-molecular-weight heparin or warfarin) should be on a stable dose.
   5. AST or ALT ≤3 x ULN. Patients with liver metastases must have AST and ALT ≤5.0 x ULN.
   6. Total bilirubin <2 mg/dL. Patients with Gilbert's Syndrome must have a total bilirubin ≤3.0 mg/dL.
   7. Serum creatinine <1.5 mg/dL or measured creatinine clearance ≥50 ml/min calculated using the Cockcroft-Gault glomerular filtration rate estimation: (140 - age) × (weight in kg) × (0.85 if female)/72 × (serum creatinine in mg/dL).
9. Patients with documented LVEF of ≥ 45%.
10. Patients with documented FEV1, FVC and DLCO ≥ 50% tested by a pulmonary function test.
11. Patients must be seronegative for HIV antibody (patients who are HIV seropositive may be less responsive and more susceptible to toxicities related to this experimental treatment since they may have a decreased immune competence).
12. Patients must be seronegative for active hepatitis B (defined as having a negative hepatitis B surface antigen [HBsAg] test), and seronegative for hepatitis C antibody. Patients with a history of hepatitis B virus (HBV) infection and having a negative HBsAg test and a positive antibody to hepatitis B surface antigen (HBsAg) are eligible. Patients with the hepatitis C antibody test positive are eligible only if tested for the presence of antigen by RT-PCR and be HCV RNA negative.
13. Life expectancy ≥3 months.
14. Patients who are of childbearing potential (postmenarcheal who has not reached a postmenopausal state and has not undergone surgical sterilization) or have partners of childbearing potential must agree to use a highly effective method of contraception during the study and for at least 6 months after the last dose of IL-2.
15. Female participants: a female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Women of non-childbearing potential (WONCBP).
    2. Women of childbearing potential (WOCBP), who:

    i. Agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year from screening until 6 months after the infusion of the TIL product. Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal occlusion, male sterilization, and copper intrauterine devices.

    ii. Have a negative pregnancy test (blood) within one week before the first study treatment administration (applicable to premenopausal women and women ≤2 years after the start of menopause (menopause is defined as amenorrhea for <2 years).

    iii. Refrain for donating ovules during the study
16. Male Participants: during the treatment period and for at least 2 months after the last dose of study treatment, agreement to:

    1. Remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures such as a condom or a contraceptive method that result in a failure rate of <1% per year, with partners who are WOCBP.
    2. Refrain from donating sperm during the study.
    3. Inform if his partner gets pregnant during this time.
17. Any toxicity related to prior systemic therapy must have recovered to grade 1 or less according to NCI-CTCAE v5.0 at least 4 weeks before enrollment, except for alopecia, vitiligo, or endocrinopathy managed with replacement therapy, and Grade ≤2 peripheral neuropathy.

    Note: Other Grade 2 AEs that are deemed clinically insignificant by treating physician and in consultation with Medical Monitor are permitted.
18. Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.

Exclusion Criteria:

1. Patients with more than two brain metastases. Note: Patients with brain metastases > 1cm in diameter or perilesional edema on MRI scan must be definitively-treated and stable for at least 4 weeks, and the patient must not require corticosteroid treatment >10 mg prednisone or equivalent per day to be considered for enrollment;
2. Patients with symptomatic brain metastasis.
3. Patients with leptomeningeal carcinomatosis.
4. Patients with an active concurrent or history within the past 3 years of invasive malignancy, except for non-melanoma skin cancer, cervical and bladder carcinoma in situ, good prognosis ductal carcinoma in situ of the breast, or prostate carcinoma that is in remission under androgen deprivation therapy for >2 years. Other exceptions may apply and require discussion between the Investigator and the Medical Monitor.
5. Patients with an active systemic infection requiring anti-infective treatment within 14 days before preparative lymphodepleting therapy.
6. Patients with active hepatitis B or hepatitis C.
7. Patients with active autoimmune disease requiring immunosuppressive treatments.
8. Patients with a history of organ or bone marrow transplantation.
9. Patients with any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and AIDS).
10. Patients requiring regular treatment with steroids at a dose higher than prednisone 10 mg/day (or equivalent).

    Note: use of inhaled, topical steroids and use of systemic physiologic corticosteroid replacement therapy are permitted.
11. Patients with current or history within the last 6 months, as determined by the Investigator, of clinically significant, progressive, and/or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac, gastroenterological or neurological disease.
12. Patients with a history of coronary revascularization or ischemic symptoms within 6 months of first dose of NMA-LD chemotherapy.
13. History of idiopathic pulmonary fibrosis or evidence of active pneumonitis (any origin).
14. Patients with allergies to any of the compounds included in any of the treatment products.
15. Patients with contraindications for cyclophosphamide, fludarabine and IL-2 at per protocol doses.
16. Patients who have received any approved anti-cancer cytotoxic, anti-angiogenic and ICB therapy including radiotherapy within 4 weeks before preparative lymphodepleting therapy.

    a) Exception: palliative radiotherapy for bone metastasis >2 weeks before preparative lymphodepleting therapy, denosumab, bisphosphonates, androgen-deprivation therapy for prostate cancer and hormonal therapy for breast cancer.
17. Patients who have received any non-cytotoxic drug and molecular targeted therapy within 4 weeks before preparative lymphodepleting therapy (or within five half-lives of the investigational product, whichever is shorter).
18. Patients who have received any investigational agent within 4 weeks before preparative lymphodepleting therapy (or within five half-lives of the investigational product, whichever is shorter).
19. Patients who have received a live, attenuated vaccination within the 4 weeks before lymphodepleting therapy.
20. Patients who have undergone major surgery in the previous 3 weeks before lymphodepleting therapy.
21. Patients who have previously received any investigational cell or gene therapies.
22. Women of childbearing potential who are pregnant or breastfeeding.
23. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Predefined grade ≥3 relevant adverse events | During the first two weeks from the first dose of interleukin administered
  Mean number of predefined grade ≥3 relevant adverse events per treatment arm during the first two weeks from the first dose of interleukin administered. Predefined relevant adverse events are rash, fatigue, myalgia, chills, fever, hypotension, arrhythmia, hypoxia, dyspnea, pulmonary distress, oliguria, edema, weight gain, diarrhea, confusion, headache, anxiety, ALT increase, AST increase, bilirubin increase, and serum creatinine increase according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
PRO CTCAE | From the baseline assessment (within 3 days before TIL infusion) to the first post-treatment evaluation (at week 6 after TIL infusion).
  Change of PRO CTCAE composite score (score 0-3 for each symptom) of selected events (diarrhea, fatigue, shortness of breath, rash, swelling, chills, heart palpitations, insomnia, anxious, sad, headache and muscle pain) from the baseline assessment (within 3 days before TIL infusion) to the first post-treatment evaluation.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | From lymphodepleting chemotherapy start through 30 days after the last dose of IL-2, or until the first dose of the subsequent anti-cancer therapy, whichever occurs first.
  Nature, frequency, and severity of treatment related adverse events according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) per treatment arm.
Overall Response Rate (ORR) | From the date of baseline until the date of disease progression, assessed up to 60 months.
  Overall Response Rate (ORR) per RECIST v1.1 as assessed by investigator.
Duration of Response (DOR) | From the time measurement criteria are met for CR or PR until the first date that recurrent or progressive disease is objectively documented, assessed up to 60 months.
  Duration of Response (DOR) per RECIST v1.1 as assessed by investigator.
Percentage change of tumor size | From the date of baseline until the date of best response, assessed up to 60 months.
  Tumor size calculated as the percentage change
Progression Free Survival (PFS) | From the date of baseline until the date of disease progression, assessed up to 60 months.
  Progression Free Survival (PFS) is defined as the time from the date of treatment administration to the date of first documentation of disease progression or death due to any cause, whichever occurs first. For a patient who has not progressed and is last known to be alive, PFS will be censored at the last response assessment that is stable disease (SD) or better.
Overall survival (OS) | From the date of treatment administration to the date of death, assessed up to 60 months.
  Overall survival (OS) defined from the date of treatment administration to the date of death.
Use of Hospital Anxiety and Depression Scale (HADS) | From the date of baseline (within 3 days before TIL infusion) to sixth month during post-hospitalization follow-up (within 8 weeks after the planned visit)
  Patient reported Anxiey and Depression as measured by the "Hospital Anxiety and Depression Scale" (HADS).
  HADS evaluates the symptoms of anxiety and depression. It is composed of two subscales: Depression and Anxiety, each with seven items. The score for each subscale can change from 0 to 21, since each item has four options as answers, ranging from absence/minimal presence = 0, to maximum presence = 3. The higher the score obtained, the greater the intensity or severity of the symptoms. The period in which the patient is examined corresponds to the last seven days.
Qualitative interviews of patient experience | At clinical visit before the first CT scan of response evaluation (approximately 6 weeks after the beginning of treatment)
  Qualitative evaluation of patient experience regarding themes around the care journey, expectations and uncertainty whilst undergoing TILs therapy through in-person or virtual qualitative interviews conducted before disease re-evaluation
Costs of TIL-ACT using HD-IL-2 and ANV419 | From first patient who has started study treatment until the last subject's last study-related phone call or visit, assessed up to 60 months.
  Direct and indirect costs of TIL-ACT using HD-IL-2 and ANV419.
Quality of life questionnaire (EORTC QLQ-C30) | From baseline (within 3 days before TIL infusion) to sixth month during post-hospitalization follow-up (within 8 weeks after the planned visit)
  Trajectories of quality of life and symptomatology using the EORTC QLQ-C30 questionnaire.
Quality of life questionnaire (EQ-5D-5L) | From baseline (within 3 days before TIL infusion) to sixth month during post-hospitalization follow-up (within 8 weeks after the planned visit)
  Trajectories of quality of life and symptomatology using the EQ-5D-5L questionnaire.
Capture of physiological parameters (Heartbeat) | From baseline (within 3 days before TIL infusion) to sixth month during post-hospitalization follow-up (within 8 weeks after the planned visit)
  Rate of heartbeat (beats per minute (bpm)) using wearable device (Garmin VivoSmart 5 smartwatch).
Capture of physiological parameters (Mobility) | From baseline (within 3 days before TIL infusion) to sixth month during post-hospitalization follow-up (within 8 weeks after the planned visit)
  Mobility capture (in kms) by wearable device (Garmin VivoSmart 5 smartwatch).
Capture of physiological parameters (SpO2) | From baseline (within 3 days before TIL infusion) to sixth month during post-hospitalization follow-up (within 8 weeks after the planned visit)
  SpO2 percentage amount (in %) using wearable device (Garmin VivoSmart 5 smartwatch).
Capture of physiological parameters (Sleep cycle) | From baseline (within 3 days before TIL infusion) to sixth month during post-hospitalization follow-up (within 8 weeks after the planned visit)
  Capture of sleep cycle by wearable device (Garmin VivoSmart 5 smartwatch). It measures how long the most important phases of sleep lasted: light, deep and REM, as well as the moments at which each phase occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Garralda, Principal Investigator — Vall d'Hebron Institute of Oncology
Locations (1):
- Vall d'Hebron Institute of Oncology, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No